CLINICAL TRIAL: NCT02959489
Title: Risk Evaluation and Education for Alzheimer's Disease - the Study of Communicating Amyloid Neuroimaging (REVEAL-SCAN)
Acronym: REVEAL-SCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of Pennsylvania (Other); University of Michigan (Other); Duke University (Other); Boston University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Robert C. Green, MD, MPH, Principal Investigator of REVEAL-SCAN, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: RF1AG047866 (NIH); 1RF1AG047866-01A1 (NIH)
Record Dates: First submitted 2016-10-24; First posted 2016-11-09 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease; Amyloid Beta-Peptides; Risk Assessment; Education; Neuropsychological Tests; Neuroimaging
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amyloid Brain Imaging Non-Disclosure (Active Comparator): Subjects will receive their Alzheimer's disease (AD) risk assessment based on age, gender, family history and ancestry.
  Interventions: Behavioral: Alzheimer's Disease Risk Disclosure
- Amyloid Brain Imaging Disclosure (Experimental): Subjects will receive both their "elevated" or "not elevated" amyloid neuroimaging results based on their brain scan interpretation and Alzheimer's disease (AD) risk disclosure. The AD risk assessment is based on age, gender, family history and ancestry.
  Interventions: Behavioral: Amyloid Brain Imaging and Alzheimer's Disease Risk Disclosure

INTERVENTIONS:
Behavioral: Alzheimer's Disease Risk Disclosure — Subjects will learn a numerical risk estimate for the chance of progressing to dementia of the Alzheimer's type.
  Arms: Amyloid Brain Imaging Non-Disclosure
Behavioral: Amyloid Brain Imaging and Alzheimer's Disease Risk Disclosure — Subjects will learn their own "elevated" or "not elevated" amyloid results and a numerical risk estimate for the chance of progressing to dementia of the Alzheimer's type.
  Arms: Amyloid Brain Imaging Disclosure

SUMMARY:
This study is intended to examine the impact of learning amyloid brain imaging results among asymptomatic older adults, and how to safely communicate these results and educate on the risk of developing Alzheimer's disease.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a brain disease and is the most common form of dementia. Clinical trials for the prevention of AD have been moving to enroll subjects at increasingly earlier time-points, and are now focusing upon individuals who are not only cognitively normal but also have biomarkers associated with an increased risk of developing AD. Detecting one specific biomarker on brain scans, i.e. amyloid-beta protein, is currently used to inform diagnoses in cognitively impaired individuals, and its use may expand to pre-clinical AD cases as preventive therapies are developed.

In the REVEAL-SCAN clinical trial, the investigators are examining the psychological and behavioral impact of learning "elevated" and "not elevated" amyloid neuroimaging results pertaining to the risk of progressing to Alzheimer's disease dementia by age 85 among cognitively normal older adults. The study's goal is to learn how to communicate these amyloid brain scan results and the risk of developing AD dementia by age 85 in a diverse population of cognitively normal older adults. Findings will be relevant to future decision-making in research trials and clinical practices.

Study sites will enroll older, cognitively normal individuals (approx. 370 total) using APOE genotyping to enrich the enrollment sample such that roughly 100 of those scanned will have elevated amyloid brain scan results. From this enriched sample, participants (approximately 25% African-American) will all receive their Alzheimer's Disease Dementia Risk Assessment based on known risk factors. Half of the participants will be randomized to also learn their amyloid brain scan result at that time, while the other half will learn their scan result 6 months later. Cognitive, psychological, and behavioral outcomes will be compared between these two groups. Participants will be followed for up to 9 months with up to 7 in-person visits and 5 phone calls.

REVEAL-SCAN is the first multisite randomized clinical trial to explore the benefits, risks and limitations of disclosing amyloid results, and will help researchers and clinicians understand downstream implications of this emerging technology as it becomes increasingly utilized to compile comprehensive neuroimaging profiles for older adults at risk for developing Alzheimer's disease dementia.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking individuals (65-80 years old) with normal cognition
* Individuals with at least one first-degree relative with Alzheimer's disease (parent, sibling, child)
* Individuals who have a close friend, relative or spouse (18+) willing to be a study partner. Study partners complete surveys and interviews, accompany the study subject to the second in-person study visit, and may be asked to attend other/all study visits.
* Individuals who are willing to give a cheek swab sample to undergo blinded (undisclosed) APOE genotyping
* Individuals willing to participate in a randomized clinical trial of amyloid imaging disclosure

Exclusion Criteria:

* Individuals who have suffered from a stroke or head trauma
* Individuals who have active medical or psychiatric illness that is unstable or progressive
* Individuals who are taking acetylcholinesterase inhibitors of memantine

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 315 (Actual)
Dates: Start 2016-11; Primary Completion 2020-05-13 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Change in baseline neuropsychological performance compared to 6 weeks and 6 months post-disclosure | Baseline, 6 weeks post-disclosure, 6-months post-disclosure
  Assessed via the A4 Study's Preclinical Alzheimer Cognitive Composite (ADCS-PACC) battery, which combines tests that measure episodic memory, timed executive function, and global cognition.

SECONDARY OUTCOMES:
Change in baseline measure scores on scales and questionnaires of psychological distress compared to 6 weeks and 6 months post-disclosure. | Baseline, 6 weeks post-disclosure, 6-months post-disclosure
  Psychological distress will be measured between and within participants at the same and different study time points, and will be based on participants' scores on scales and questionnaires in terms of the following related variables of psychological distress: anxiety and depression, test-specific distress, psychological impact of disclosure, quality of life, perceived time and subjective cognition.
Change in baseline measures of health behaviors compared to 6 weeks and 6 months post-disclosure to determine the type and frequency of behavior changes in response to learning risk information. | Baseline, 6 weeks post-disclosure, 6-months post-disclosure
  Assessed in participant surveys via questions evaluating: health behavior changes, advanced planning, insurance changes (i.e. purchasing or altering long-term care policies), medication changes, willingness to enroll in clinical research and tolerance of research risk.

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Green, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Jason Karlawish, MD, Principal Investigator — University of Pennsylvania; J. Scott Roberts, PhD, Principal Investigator — University of Michigan; Kathleen Welsh-Boomer, PhD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT02959489/Prot_001.pdf
  • Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT02959489/SAP_002.pdf